CLINICAL TRIAL: NCT01003886
Title: A Post Marketing Surveillance Study To Determine The Safety, Tolerability And Effectiveness Of Doxazosin Mesylate GITS Among Filipino Adult Males With Benign Prostatic Hyperplasia (BPH)
Brief Title: A Post Marketing Surveillance Study Of Doxazosin Mesylate GITS Among Filipino Patients With Benign Prostatic Hyperplasia (BPH)
Status: Completed | Type: Observational
Sponsor: Pfizer's Upjohn has merged with Mylan to form Viatris Inc. (Industry)
Responsible Party: Sponsor
Organization: Pfizer (Industry)
Other Study IDs: A0351068
Record Dates: First submitted 2009-10-28; First posted 2009-10-29 (Estimated); Results first posted 2011-10-28 (Estimated); Last update posted 2021-01-28 (Actual); Status verified 2021-01

CONDITIONS: Prostatic Hyperplasia
Keywords: post marketing surveillance Filipino benign prostatic hyperplasia BPH Doxazosin GITS
MeSH Terms: conditions — Prostatic Hyperplasia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Open Label: Adult male diagnosed with BPH and prescribed with Doxazosin mesylate GITS
  Interventions: Drug: Doxazosin mesylate GITS

INTERVENTIONS:
Drug: Doxazosin mesylate GITS — Doxazosin mesylate GITS 4mg to 8mg once daily
  Other Names: Alfadil XL

SUMMARY:
This study aims to assess the safety, tolerability and efficacy of Doxazosin GITS in Filipino patients diagnosed with Benign Prostatic Hyperplasia (BPH) under the usual clinical care setting.

DETAILED DESCRIPTION:
This is an open label study. All patients prescribed with Doxazosin GITS can be enrolled in this study.

ELIGIBILITY:
Inclusion Criteria:

* Subjects that will be included must be consistent with the approved label indication of Doxazosin mesylate GITS in the Philippines, which includes adult male diagnosed with BPH, and who are prescribed with Doxazosin mesylate GITS.

Exclusion Criteria:

* Subjects with condition that are contraindicated with Doxazosin mesylate GITS based on the approved labeling in the Philippines.

Ages: 18 Years to 90 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Filipino adult males diagnosed with Benign Prostatic Hyperplasia (BPH) and prescribed with Doxazosin mesylate GITS
Sampling Method: Non-Probability Sample
Enrollment: 989 (Actual)
Dates: Start 2009-05; Primary Completion 2011-01 (Actual); Study Completion 2011-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (60):
- Philippines (60):
  - Pfizer Investigational Site, Butuan, Agusan Del Norte
  - Pfizer Investigational Site, San Juan City, Batangas
  - Pfizer Investigational Site, Tagbilaran City, Bohol
  - Pfizer Investigational Site, Quezon City, Diliman
  - Pfizer Investigational Site, City of San Fernando, La Union
  - Pfizer Investigational Site, Ermita, Manila
  - Pfizer Investigational Site, Tondo, Manila
  - Pfizer Investigational Site, Diliman, Quezon City, National Capital Region
  - Pfizer Investigational Site, Pasig, National Capital Region
  - Pfizer Investigational Site, Angeles City, Pampanga
  - Pfizer Investigational Site, Angeles
  - Pfizer Investigational Site, Angeles City
  - Pfizer Investigational Site, Bacolod City
  - Pfizer Investigational Site, Baguio City
  - Pfizer Investigational Site, Bohol
  - Pfizer Investigational Site, Bulacan
  - Pfizer Investigational Site, Butuan
  - Pfizer Investigational Site, Cagayan de Oro
  - Pfizer Investigational Site, Cebu
  - Pfizer Investigational Site, Cebu City
  - Pfizer Investigational Site, City of Muntinlupa
  - Pfizer Investigational Site, Davao City
  - Pfizer Investigational Site, Gallares City
  - Pfizer Investigational Site, General Santos
  - Pfizer Investigational Site, Iligan City
  - Pfizer Investigational Site, Ilocos Norte
  - Pfizer Investigational Site, Kalibo
  - Pfizer Investigational Site, Kalibo Aklan
  - Pfizer Investigational Site, La Union
  - Pfizer Investigational Site, Laguna
  - Pfizer Investigational Site, Laoag
  - Pfizer Investigational Site, Lingayen, Pangasinan
  - Pfizer Investigational Site, Makati City
  - Pfizer Investigational Site, Malabon
  - Pfizer Investigational Site, Manadaluyong
  - Pfizer Investigational Site, Mandaluyong
  - Pfizer Investigational Site, Mandaue City
  - Pfizer Investigational Site, Manila
  - Pfizer Investigational Site, Marikina City
  - Pfizer Investigational Site, Mindanaw
  - Pfizer Investigational Site, Nueva Ecija
  - Pfizer Investigational Site, Nueva Vizcaya
  - Pfizer Investigational Site, Ozamiz
  - Pfizer Investigational Site, Pampanga
  - Pfizer Investigational Site, Pasig
  - Pfizer Investigational Site, Philippines
  - Pfizer Investigational Site, Quezon
  - Pfizer Investigational Site, Quezon City
  - Pfizer Investigational Site, Rizal
  - Pfizer Investigational Site, San Jose
  - Pfizer Investigational Site, Surigao City
  - Pfizer Investigational Site, Tacloban City
  - Pfizer Investigational Site, Tagbilaran City
  - Pfizer Investigational Site, Tagum
  - Pfizer Investigational Site, Tarlac City
  - Pfizer Investigational Site, Tuguegarao City
  - Pfizer Investigational Site, Valenzuela
  - Pfizer Investigational Site, Vigan
  - Pfizer Investigational Site, Visayas
  - Pfizer Investigational Site, West Fairview, Quezon City

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A0351068&StudyName=A%20Post%20Marketing%20Surveillance%20Study%20Of%20Doxazosin%20Mesylate%20GITS%20Among%20Filipino%20Patients%20With%20Benign%20Prostatic%20Hyperplasia%20%28BPH%29

RESULTS

PARTICIPANT FLOW:
Groups:
- Doxazosin GITS: Doxazosin mesylate gastrointestinal therapeutic system (GITS) tablet taken orally at a dose of 4 milligram (mg) once daily (QD) or 8 mg QD for 12 weeks.
Period: Overall Study
Arm/Group | Doxazosin GITS
Started | 989
Completed | 759
Not Completed | 230
Not completed — Lack of Efficacy | 5
Not completed — Lost to Follow-up | 169
Not completed — Withdrawal by Subject | 39
Not completed — Other | 14
Not completed — Adverse Event | 3

BASELINE CHARACTERISTICS:
Arm/Group | Doxazosin GITS
Number analyzed (Participants) | 989
Age, Continuous [Mean (Standard Deviation); unit: Years] | 62.50 (10.10)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 989
Systolic blood pressure (BP) [Mean (Standard Deviation); unit: Millimeters of mercury (mmHg)] — N=900 for the parameter analyzed.
  Millimeters of mercury (mmHg) | 127.80 (15.18)
Diastolic BP [Mean (Standard Deviation); unit: mmHg] — N=900 for the parameter analyzed.
  mmHg | 80.50 (9.35)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Adverse Events (AEs)
Description: Any untoward medical occurrence in a participant who received study drug was considered an AE, without regard to possibility of causal relationship.
Time Frame: Baseline up to Week 13 (7 days after last dose)
Population: Safety population included participants who had taken at least 1 dose of the study medication.
Measure: Number; unit: Participants
Arm/Group | Doxazosin GITS
Number analyzed (Participants) | 989
Participants | 14

2. Secondary Outcome: Percent Change From Baseline in the International Prostate Symptom (IPSS) Total Score at Week 4 and Week 12
Description: The IPSS total score is obtained by combining the scores of the responses to 1 through 7 component questions all of which were on a 6 point likert scale. Each question is scored from 0-5 for an IPSS range of 0-35 points where 0 = best possible score to 35 = worst possible score.
Time Frame: Baseline, Week 4 and Week 12
Population: Full analysis set (FAS) population included participants who had taken at least 1 dose of the study medication. Missing post-baseline data was replaced by the last observation carried forward (LOCF). The 'n' is signifying those participants who received study drug and were evaluated for this measure at the time points for each group respectively.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Doxazosin GITS
Number analyzed (Participants) | 989
Units on a scale
  Baseline (n=962) | 22.30 (6.87)
  Percent change at Week 4 (n=889) | -44.90 (23.14)
  Percent change at Week 12 (n=637) | -65.10 (23.96)
  Percent change at Week 12 (LOCF) (n=934) | -61.40 (24.66)

3. Secondary Outcome: Percent Change From Baseline in the IPSS Quality of Life (QoL) Score at Week 4 and Week 12
Description: The IPSS QoL Score is obtained by assessment of a single QoL question on a 7-point likert scale which was scored on a scale of 0-6 where 0 = best possible score to 6 = worst possible score.
Time Frame: Baseline, Week 4 and Week 12
Population: FAS population included participants who had taken at least 1 dose of the study medication. Missing post-baseline data was replaced by the LOCF. The 'n' is signifying those participants who received study drug and were evaluated for this measure at the time points for each group respectively.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Doxazosin GITS
Number analyzed (Participants) | 989
Units on a scale
  Baseline (n=965) | 4.20 (1.04)
  Percent change at Week 4 (n=892) | -44.60 (23.62)
  Percent change at Week 12 (n=636) | -64.10 (24.08)
  Percent change at Week 12 (LOCF) (n=936) | -60.50 (25.37)

4. Secondary Outcome: Change From Baseline in Systolic BP at Week 4 and Week 12
Description: Values at Week 4 and Week 12 minus value at baseline.
Time Frame: Baseline through Week 12
Population: Safety population included participants who had taken at least 1 dose of the study medication. The 'n' is signifying those participants who received study drug and were evaluated for this measure at the time points for each group respectively.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Doxazosin GITS
Number analyzed (Participants) | 989
mmHg
  Change at Week 4 (n=816) | -3.80 (11.07)
  Change at Week 12 (n=583) | -5.70 (11.22)

5. Secondary Outcome: Change From Baseline in Diastolic BP at Week 4 and Week 12
Description: Values at Week 4 and Week 12 minus value at baseline.
Time Frame: Baseline through Week 12
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Doxazosin GITS
Number analyzed (Participants) | 989
mmHg
  Change at Week 4 (n=816) | -1.50 (7.95)
  Change at Week 12 (n=583) | -2.40 (8.49)

6. Secondary Outcome: Percentage of Participants With Postural Hypotension
Description: Postural or orthostatic hypotension is a medical condition where blood pressure falls rapidly after the body changes position most commonly occurring after standing up after sitting for long periods of time.
Time Frame: Baseline up to Week 13 (7 days after last dose)
Population: Safety population included participants who had taken at least 1 dose of the study medication.
Measure: Number; unit: Percentage of participants
Arm/Group | Doxazosin GITS
Number analyzed (Participants) | 989
Percentage of participants | 0.3

ADVERSE EVENTS:
Description: The same event may appear as both an AE and a SAE. However, what is presented are distinct events. An event may be categorized as serious in one subject and as nonserious in another subject, or one subject may have experienced both a serious and nonserious event during the study.
Arm/Group | Doxazosin GITS
Serious Adverse Events (participants affected / at risk) | 0/989
Other Adverse Events (participants affected / at risk) | 14/989
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Doxazosin GITS (N=989)
Myocardial ischaemia (Cardiac disorders) | 1
Vision blurred (Eye disorders) | 1
Decreased appetite (Metabolism and nutrition disorders) | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 1
Dizziness (Nervous system disorders) | 7
Headache (Nervous system disorders) | 1
Hypertension (Vascular disorders) | 1
Hypotension (Vascular disorders) | 2
Orthostatic hypotension (Vascular disorders) | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.